CLINICAL TRIAL: NCT03597230
Title: Per-operative Exploration of the Peri-pancreatic Lymphatic Pathways During Pancreatic Surgical Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PO18091
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Resection
MeSH Terms: interventions — Coloring Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients operated on for pancreatic resection (Experimental): All consecutive patients operated on for pancreatic resection
  Interventions: Other: Dye

INTERVENTIONS:
Other: Dye — Cover key details of the intervention. Must be sufficiently detailed to distinguish between arms of a study and/or among similar interventions At the beginning of the surgical procedure, 1 ml of blue patent will be injected in the normal remaining part of the pancreas. The diffusion of the dye among all lymph node areas will be noticed by the surgeon.
  Other Names: The dye will be the blue patent, widely used for the detection of the sentinel lymph node for breast cancer

SUMMARY:
Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis (Limit : 5000 characters) Pancreatic cancer has a poor prognosis. Surgical resection is the only curative treatment. Major pancreatectomies lead to high postoperative morbidity rate, up to 30%. For some tumors, limited resection are increasedly performed, but the rate of pancreatic fistula is even higher, up to 40%.

No precise "anatomic" pancreatic segmentation currently exists. If such segmentation is described, pancreatic resections, major of minor, may have better outcomes.

The aim of this study is to demonstrate the existence of independent pancreatic segments, following the lymphatic drainage of the gland.

DETAILED DESCRIPTION:
Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures. (Limit : 32 000 characters) The prognosis and life expectancy for people with pancreatic cancer remain very low (3rd cause of mortality among all cancer). Surgical resection is the only curative treatment, whenever possible. Nevertheless, major pancreatectomies lead to high postoperative morbidity rate, in particular up to 30% fistula rate. In case of parenchyma-sparing procedures, this rate is even higher, up to 40%.

One of the reasons of these high rates might be explained by the fact that pancreatic transections are currently not performed following pancreatic segmentation. If possible, resection following vascular segmentation would prevent necrosis of the transection, resection following lymphatic segmentation would improve the lymph-node dissection, and resection following pancreatic-duct segmentation would prevent leakage from pancreatic duct stump. Nevertheless, no precise "anatomic" pancreatic segmentation currently exists.

On the other hand, the lymphatic system of the pancreas is highly complex, but the quality of the lymphadenectomy during pancreatectomy is essential since the recurrences almost always occur on the lymphatic transections. A better knowledge of the peri-pancreatic lymphatic vessels is still required.

The aim of this study is to demonstrate the existence of independent pancreatic segments, following the lymphatic drainage of the gland.

ELIGIBILITY:
Inclusion Criteria:

* All patient operated on for pancreatic resection
* Patients consenting the protocol after clear and loyal explanations

Exclusion Criteria:

* history of first abdominal surgery in the upper part
* Patients with peritoneal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-10-22 (Estimated); Study Completion 2020-10-22 (Estimated)

PRIMARY OUTCOMES:
Lymph node areas colored by the diffusion of the blue patent | 3 minutes after the injection
  At the beginning of the surgical procedure, 1 ml of blue patent will be injected in the normal remaining part of the pancreas. The diffusion of the dye among all lymph node areas will be noticed by the surgeon.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Renard Y, Perrenot C, Labrousse M, Avisse C, Rhaiem R, Piardi T, Braun M, Perez M. Exploration of peripancreatic lymphatic pathways in a live porcine model. Ann Anat. 2019 Sep;225:57-64. doi: 10.1016/j.aanat.2019.06.003. Epub 2019 Jul 5. PMID 31284072